CLINICAL TRIAL: NCT06238700
Title: Targeting Allopregnanolone to Probe Behavioral and Neurobiological Mechanisms That Underlie Depression in Women Across the Menopause Transition
Brief Title: Study on Allopregnanolone and Depression in Women Across the Menopause Transition
Acronym: SADIE-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Natalie Feldman, Psychiatrist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024P000113
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnenolone (Experimental): Participants will take 250mg of pregnenolone twice per day (daily total=500mg) for four weeks
  Interventions: Dietary Supplement: pregnenolone
- placebo (Placebo Comparator): Participants will take placebo twice per day for four weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: pregnenolone — Pregnenolone is an endogenous steroid available in the US and elsewhere as an orally administered over-the-counter supplement.
  Arms: pregnenolone
Other: placebo — Placebo pills are identical-appearing capsules containing cellulose
  Arms: placebo

SUMMARY:
This study aims to identify how enhanced allopregnanolone activity (via pregnenolone) affects behavior and neurobiology that may underlie perimenopausal depression.

DETAILED DESCRIPTION:
Midlife women are burdened with depression risk that is at least partly attributed to changing reproductive steroid dynamics across a prolonged reproductive transition. We hypothesize that declining endogenous allopregnanolone (ALLO) levels across the menopause transition underlies perimenopausal depression. This mechanistic trial aims to amplify the contrast between lower endogenous ALLO levels in perimenopausal women and higher levels induced by pregnenolone. This will be achieved by using the over-the-counter dietary supplement, pregnenolone, in a randomized, double-blind, parallel-arm, placebo-controlled trial. By manipulating ALLO levels together with key measurement of depression domains, this study harnesses the endocrine biology of perimenopause to explicate behavioral and neurobiological mechanisms underlying depression in women across the menopause transition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ages 40 to 60 years in the menopause transition
* Depressive symptoms
* Psychotropic medications are allowed if the dose is stable prior to screening and throughout the study
* Able to read Arabic numerals and perform simple arithmetic
* Able to provide written informed consent

Exclusion Criteria:

* Systemic hormone therapy
* Contraindicated medications with pregnenolone
* Systemic corticosteroid
* Other psychiatric illnesses that are considered to be primary
* Current suicidal ideation
* Active substance use disorders
* Unstable medical conditions
* Obstructive sleep apnea or other primary sleep disorders
* Abnormal hepatic and renal function
* Known allergy to progesterone, exogenous allopregnanolone, or pregnenolone
* History of head injury resulting in loss of consciousness > 20 min
* Inability to comply with barrier contraceptive methods
* Known intellectual disability
* Investigator judgement that study participation constitutes substantial risk given medical or psychiatric condition
* Current or recent participation in clinical trial expected to interfere with risk of or interpretation of study data
* Inability to comply with study procedures

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Within-person change in score on the Ruminative Responses Scale | Baseline to 2 weeks
  The Ruminative Responses Scale (RRS) comprises 22 items which ask how frequently the participant thinks certain statements when they feel depressed. Each item is scored from 1-4. Total scores range from 22-88 with higher scores indicating more severe rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD MSc, Principal Investigator — Brigham and Women's Hospital; Katherine Burdick, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No